CLINICAL TRIAL: NCT04795362
Title: S100B Kinetic During the Occurrence and Treatment of Delayed Cerebral Ischaemia After a Subarachnoid Haemorrhage.
Acronym: SKinDCI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1081; 2021-A00048-33 (Other: ID-RCB)
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-04

CONDITIONS: Subarachnoid Hemorrhage
Keywords: subarachnoid haemorrhage; S100B; Delayed cerebral ischemia
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with Delayed cerebral ischemia: 50 adult patients hospitalized in neurological intensive care unit for subarachnoid hemorrhage, in whom the onset of delayed cerebral ischemia is suspected will be included.
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — 5 tubes of 1 milliliters (ml) will be sampled on a catheter placed as part of the usual practice every hour for 4 hours (at Time 0, at Time 1 hour, at time 2hours, at Time 3 hours, at time 4 hours) as soon as DCI is suspected.
  In the event of a mechanical angioplasty decision, the samples will be continued (Time 0, Time 2 hours, Time 4 hours, Time 6hours, Time 12 hours, Time 24 hours, so 6 samples of 1 ml).

SUMMARY:
Nearly half of the survivors of subarachnoid haemorrhage (SAH) retain irreversible neurological damage resulting from the early lesions associated with the initial bleeding, and the occurrence of possible delayed cerebral ischaemia (DCI). The early diagnosis of the occurrence of an DCI is therefore a major challenge in order to optimise management before irreversible lesions are formed. However, the means of diagnosis are often not available, and up to a third of DCI are discovered on follow-up images when the lesions are already present. Among the markers of brain injury, S100 calcium-binding protein B (S100B) is an astrocyte protein released into the bloodstream at the time of the appearance of a brain lesion. Its short half-life makes it a prime candidate for patient follow-up to diagnose a new ischemic lesion and assess the effectiveness of its management.

Among the elements at the origin of DCI, the occurrence of proximal vasospasm is the main element on which we can have a therapeutic action. The strategy implemented in the department consists of performing a mechanical angioplasty when proximal vasospasm is detected with a decrease in downstream cerebral perfusion. Nevertheless the benefit of this therapeutic action is discussed and there is currently no early marker of the effectiveness of this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Patient hospitalised in the neurological intensive care unit for a subarachnoid haemorrhage.
* Delayed cerebral ischaemia suspected during routine care.
* Presence of a catheter (arterial or venous) for repeated sampling.
* Patient having been informed and having formulated his non-opposition or close to the patient having been informed and having formulated his non-opposition. In this case, the patient's non-opposition will be collected as soon as his condition allows it.

Exclusion Criteria:

* Pregnant or breastfeeding women in class.
* Patients under legal protection, guardianship, curatorship, under judicial safeguard.
* Patients participating in a study that may interfere with this study.
* Persons under psychiatric care under duress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized in neurological intensive care unit for subarachnoid hemorrhage, in whom the onset of delayed cerebral ischemia is suspected will be included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
S100B serum concentration after DCI suspicion. | through study completion, an average of 2 year
  S100B repeated samples, measure with an ELISA kit from ROCHE diagnostic.
  Measurement of the evolution of the S100B during at T0, T1h, T2h, T3h, T4h after the suspicion of DCI by the physician in charge.
  If an intravascular angioplasty procedure is performed S100B kinetic will be measured at T0, T2h, T4h, T6h, T12h and T24h after the procedure.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Femme Mère Enfant, Bron
  - Hôpital Gabriel Montpied, Clermont-Ferrand